CLINICAL TRIAL: NCT01844427
Title: Memantine Monotherapy for Executive Dysfunction and ADHD: A Pilot Study
Brief Title: Memantine Monotherapy for Executive Dysfunction and ADHD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013P000520
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: ADHD; Executive Function Deficits (EFD's)
Keywords: ADHD; Executive function deficits; Psychiatry; Psychopharmacology; Namenda
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memantine HCl (Active Comparator): Memantine administered in capsule form twice daily for 12 weeks and titrated up to a maximum daily dose of 20mg.
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): Masked placebo administered in capsule form twice daily for 12 weeks. Placebo titration will be titrated according to the same procedure as active memantine.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Memantine HCl is an NMDA antagonist currently FDA approved for the treatment of moderate to severe Alzheimer's-type dementia.
  Other Names: Namenda
  Arms: Memantine HCl
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a 12-week clinical trial evaluating the efficacy and safety of memantine hydrochloride (Memantine HC1, brand name Namenda) in the treatment of executive function deficits (EFDs) in adults with Attention Deficit Hyperactivity Disorder (ADHD). After screening procedures, memantine is prescribed in randomized, double-blind fashion (equal chance of medication or placebo) for 12 weeks.

The investigators hypothesize that memantine hydrochloride will prove to be an effective, safe, and well-tolerated agent for the treatment of EFDs in individuals with ADHD interested in non-stimulant medications.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults ages 18-45 years;
2. a diagnosis of DSM-IV [78] ADHD-combined type
3. a score of at least 20 on the AISRS (a score of 20 in the AISRS identifies subjects with at least moderate severity of symptoms);
4. a BRIEF-A Global Executive Composite T-score of >6; and
5. proficiency in English. -

Exclusion Criteria:

1) Pregnant or nursing females; 2) investigator and his/her immediate family (spouse, parent, child, grandparent, or grandchild); 3) any serious, unstable medical illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease and hypertension), endocrinologic, neurologic, immunologic, or hematologic disease; 4) hypersensitivity to memantine; 5) multiple adverse drug reactions; 6) current or past history of seizures; 7) any history of a major psychiatric disorder including schizophrenia, psychosis, bipolar disorder (BPD), or autism spectrum disorder (ASD); 8) meets DSM-IV criteria in the last month for major depression or any major anxiety disorder or has a Hamilton Rating Scale for Anxiety (HAM-A) or Hamilton Rating Scale for Depression (HAM-D) score greater than 14; 9) meets DSM-IV criteria for substance abuse or dependence in the last month or has a positive drug urine screen; 10) judged to be at serious suicidal risk; 11) use of any other concomitant medication with primarily central nervous system activity; or 12) IQ < 80.

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Brief-A Self-Report | Baseline to 12 weeks